CLINICAL TRIAL: NCT04819594
Title: The Effects of Aromatherapy on the Stress Levels of Nurses Working in an Urban, Safety-Net Community Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Justin Buchert, Quality Specialist, Parkland Health and Hospital System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU-2020-1413
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Stress Levels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Nurses will wear the Elequil aromatabs ® (100% pure essential oil) over a four-hour period
  Interventions: Other: Elequil aromatabs ®

INTERVENTIONS:
Other: Elequil aromatabs ® — 100% pure essential oils in a unique controlled delivery system for relaxation, comfort, and sleep. Scented tabs on a self-adhesive label will be placed on the nurses's uniform for 4 hours to provide aromatherapy for the clinical setting.

SUMMARY:
Parkland Hospital inpatient nursing staff will be the focus of this study. This project aims to investigate the use of lavender on the stress levels associated with the nursing role. Nurses will wear the Elequil aromatabs ® over a four-hour period and a post survey will be given to assess root cause of stress and changes related to intervention.

DETAILED DESCRIPTION:
Nurses today are facing unprecedented patient acuities, burnout, fear, uncertainty, a continuously evolving workflow and nursing shortages, Therefore, workplace-related stress has become one of today's most serious occupational hazards. Aromatherapy can be a convenient, inexpensive, and non-invasive method of stress relief. There is little research regarding the efficacy of aromatherapy by means of inhaling essential oils in reducing workplace stress-related symptoms among nurses. Therefore, this study will examine the efficacy of lavender-scented aromatherapy tabs (Elequil ® aromatabs ®) in reducing job stress-related symptoms among nurses.

The study for the participants goes as follows:

1. Nurse identified by:

   * Leadership
   * Self-identified
   * SPARKS member
2. Process:

   * Identified nurse will be informed and consented regarding the study.
   * An aromatab will be given to the nurse.
   * They will place the aromatab on their uniform top to allow for continuous exposure to the scent.
   * Four (4) hours later - nurse completes survey as to the effects of the aromatab
   * Completed survey is placed in research file at charge nurse desk in opaque folder.

Data to be used within the research project will be obtained from the collected survey forms.

Recruitment will be completed face-to-face between the SPARKS team member, leadership, or self -identification of the potential subject. Considerable care will be taken so that the person contacted does not feel pressured to participate.

The research team will meet prior to enrolling the first participant, during and upon completion of data collection. Any safety concerns will be addressed at those times. At any time during data collection, the PI's or any study team members may request that the team meets to address a safety concern. Study participants will be assured of anonymity and confidentiality of the data and they will also be reminded that they can withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Nurses volunteering to participate in the study and are experiencing stress while at work

Exclusion Criteria:

* Known allergies or sensitivities to aromatherapy products, a history of respiratory problems, asthma, allergies to fragrance, or lost sense of smell. Those nurses who have had serious disease complications will also be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Mean change in stress levels as measured by Nurse Survey | Baseline, 4 hours post intervention (aromatherapy)
  Nurse Survey is used for measuring the level of stress in nurses who agree that the intervention reduced their stress levels. Possible scores range from 0 - 10 with higher scores indicating severe stress levels (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Justin Buchert, MSN, M.Ed., MS, RN, Principal Investigator — Parkland Health and Hospital System
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No